CLINICAL TRIAL: NCT07167199
Title: Subcuticular Absorbable Staples Versus Conventional Skin Closure in Women Undergoing Cesarean Delivery: A Randomized Control Trial
Brief Title: Absorbable Staples Versus Conventional Skin Closure in Women Undergoing Cesarean Delivery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: INOVA-2024-333
Record Dates: First submitted 2025-08-26; First posted 2025-09-11 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy

STUDY DESIGN:
Intervention Model Description: Subjects who agree to participate in the study will be randomized to one of the two groups below in a 1/1 allocation
Who Masked: Outcomes Assessor
Masking Description: Reviewers of wound cosmetics during the post operative time will be blind to the intervention. However, surgeon at the time skin closure and patient will not be blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Suture wound closure (Active Comparator): Absorbable Moncryl sutures for closure of cesarean skin incision
  Interventions: Procedure: Subcuticular monocryl suture
- Absorbable staple wound closure (Experimental): Staples will be applied as per the manufacturer's instructions intraoperatively using INSORB device manufactured by CooperSurgical.
  Interventions: Device: Subcuticular absorbable staple using Insorb device

INTERVENTIONS:
Procedure: Subcuticular monocryl suture — Under the skin suture placed by hand
  Arms: Suture wound closure
Device: Subcuticular absorbable staple using Insorb device — Under the skin stapling device that delivers absorbable staples
  Arms: Absorbable staple wound closure

SUMMARY:
Despite the high numbers of cesareans being performed, scientific evidence behind which surgical techniques are best remains uncertain. Our objective is to determine if subcuticular absorbable staples improve operative time and wound cosmetics

DETAILED DESCRIPTION:
This will be an open-label randomized controlled clinical trial. Women undergoing cesarean delivery will be randomized to have either standard wound closure with Monocryl suture or absorbable subcuticular staples placed by INSORB skin stapling device. The INSORB under the skin stapling device is FDA approved but not currently used as standard of care at Inova. We will exclude women with intraamniotic infection, immunosuppression, active skin infection, those unlikely to be followed-up after delivery, or unable to provide consent.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Women ≥ 24 weeks viable gestation
* Will be undergoing cesarean delivery

Exclusion Criteria:

* Patient unwilling or unable to provide consent.
* No or very limited prenatal care or a non-resident patient who is unlikely to follow-up after delivery.
* Immunosuppressed subjects: i.e., taking systemic immunosuppressant or steroids (e.g. transplant subjects; not including steroids for lung maturity), HIV with CD4 <200, or other
* Decision not to have skin closure (e.g. secondary wound closure, mesh closure)
* Current skin infection
* Coagulopathy
* High likelihood of additional surgical procedure beyond cesarean (e.g. scheduled hysterectomy, tubal ligation, bowel or adnexal surgery)
* Incarcerated individuals
* Intraamniotic infection
* Subjects participating on other treatment trials or studies that would interfere with the current study's primary outcome.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 237 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Operating time | Time from the start of surgery through end of skin closure up to 8 hours
  Total time for the procedure

SECONDARY OUTCOMES:
Wound Cosmesis | Up to six weeks post partum
  A digital photograph of the incision will be obtained on wound check visit POD 5-10 days and 4-6 weeks post partum. Each photograph will be evaluated by independent blinded research staff using the Stony Brook Scar Evaluation Scale. These scores are totaled to obtain the final score. The Stony Brook Scar Evaluation will score the scar from 0-5 where 5 shows significant healing.
Post Operative Pain | up to 3 days post-operatively
  Analog pain scale ranging from 0-10. This is a standard question that nurses as during the post partum period while in the hospital and clinic/nursing visits. The numerical score will be recorded from the patient's chart.
  A score of 0 means no pain, and 10 means the worst pain.

OTHER OUTCOMES:
Number of Adverse Events | Up to 6 weeks post-partum
  Allergic reactions: anaphylaxis, angioedema, skin rashes, including Stevens Johnson and Toxic Epidermal Necrolysis
Number of participants with any unscheduled postpartum visit | up to 30 days post-operatively
  Any additional postpartum clinic appointments for medical or clinical concerns beyond the routinely scheduled visits. Participants are counted once, regardless of number or type of visits
Skin Closure Time in Minutes | Time from start of skin closure to end of skin closure up to 2 hours
  Minutes it takes for closure of the skin at time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Saad, MD, Principal Investigator — Inova Fairfax Medical Center
Locations (1):
- Inova Fairfax Medical Campus, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: No